CLINICAL TRIAL: NCT03127631
Title: The Role of Androgen Deprivation Therapy In Cardiovascular Disease - A Longitudinal Prostate Cancer Study (RADICAL PC1) & A RAndomizeD Intervention for Cardiovascular and Lifestyle Risk Factors in Prostate Cancer Patients (RADICAL PC2)
Brief Title: A RAndomizeD Intervention for Cardiovascular and Lifestyle Risk Factors in Prostate Cancer Patients
Acronym: RADICALPC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Prostate Cancer Canada (Other); Canadian Cancer Society (CCS) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: RADICALPC_009-001
Record Dates: First submitted 2016-09-07; First posted 2017-04-25 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer; Cardiovascular Disease
Keywords: Androgen Deprivation Therapy
MeSH Terms: conditions — Prostatic Neoplasms; Cardiovascular Diseases | interventions — Nutritional Status; Exercise; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Simvastatin; Atorvastatin; Rosuvastatin Calcium; Pravastatin; Angiotensin-Converting Enzyme Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (2):
- Randomized - Intervention (Active Comparator): The intervention will consist of a systematic cardiovascular and lifestyle risk factor modification strategy, including dietary and exercise advice, advice to quit smoking, and the prescription of open-label statins, ACE-I, and other antihypertensive medications where appropriate.
  Interventions: Behavioral: Nutrition; Behavioral: Exercise; Behavioral: Smoking cessation; Drug: Statin (such as Simvastatin, Atorvastatin, Rosuvastatin, Pravastatin); Drug: ACE inhibitor
- Randomized - Control (No Intervention): The control will consist of usual clinical care, which may include a referral to a cardiologist or internist, or the use of treatments included in the intervention as clinically indicated, if part of the treating physician's standard practice.

INTERVENTIONS:
Behavioral: Nutrition — Standardized advice on healthy diet practices.
  Arms: Randomized - Intervention
Behavioral: Exercise — Standardized advice on exercise including strength training and resistance training exercises.
  Arms: Randomized - Intervention
Behavioral: Smoking cessation — Advice to quit smoking, if applicable, and on available aids to quit smoking,
  Arms: Randomized - Intervention
Drug: Statin (such as Simvastatin, Atorvastatin, Rosuvastatin, Pravastatin) — Prescription for a low to moderate dose statin, such as simvastatin 10-40mg daily, atorvastatin 10-40mg daily, rosuvastatin 5-20mg daily or pravastatin 10-40mg daily.
  Arms: Randomized - Intervention
Drug: ACE inhibitor — Prescription for an ACE-I (preferable) or an angiotensin receptor blocker for baseline systolic blood pressure greater >130mmHg, or other blood pressure lowering medication as applicable.
  Arms: Randomized - Intervention

SUMMARY:
RADICAL PC1 is a prospective cohort study of men with a new diagnosis of prostate cancer. RADICAL PC2 is a randomized, controlled trial of a systematic approach to modifying cardiovascular and lifestyle risk factors in men with a new diagnosis of prostate cancer.

DETAILED DESCRIPTION:
RADICAL PC describes two prospective studies, one of which is embedded in the other. RADICAL PC1 is a prospective cohort study of men within one year of their first diagnosis of prostate cancer, or treated with Androgen Deprivation Therapy for the first time within 6 months prior to enrollment visit, or to be treated with Androgen Deprivation Therapy for the first time within one month after the enrollment visit. Its goal will be to identify factors associated with the development of cardiovascular disease among men with prostate cancer, with a particular focus on Androgen Deprivation Therapy. RADICAL PC2 is a randomized, controlled trial embedded in RADICAL PC1. RADICAL PC2 will test a systematic approach to modifying cardiovascular and lifestyle risk factors in men within one year of their first diagnosis of prostate cancer, or treated with Androgen Deprivation Therapy for the first time within 6 months prior to enrollment visit, or to be treated with Androgen Deprivation Therapy for the first time within one month after the enrollment visit.

ELIGIBILITY:
Inclusion Criteria:

1. A man with a diagnosis of prostate cancer that is either:

* new (i.e. the diagnosis was made within 1 year of the enrolment visit) or
* treated with Androgen Deprivation Therapy for the first time within 6 months prior to the enrolment visit, or
* to be treated with Androgen Deprivation Therapy for the first time within 1 month after the enrolment visit

Exclusion Criteria:

1. Patients will be excluded if they fulfill any of the following:

   1. are unwilling to provide consent or
   2. are <45 years of age, or
   3. prostate cancer was found incidentally following cystectomy for bladder cancer
2. Patients will be eligible for RADICAL PC1, but will not be eligible for RADICAL PC2 if they:

   1. see a cardiologist every year, or
   2. both take a statin and have systolic blood pressure ≤130mmHg

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2015-10-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Outcome - Composite of Death, MI, Stroke, HF, or Arterial Revasc. | 3-5 years
  The primary efficacy outcome is the occurrence of the composite of cardiovascular death, myocardial infarction, stroke, heart failure, or arterial revascularization.

SECONDARY OUTCOMES:
Secondary Efficacy Outcome - Composite of Death, MI, Stroke or HF. | 3-5 years
  The occurrence of the composite of all-cause mortality, myocardial infarction, stroke, or heart failure.
Secondary Efficacy Outcome - Composite of Death, MI, Stroke | 3-5 years
  The composite of cardiovascular death, myocardial infarction, or stroke.
Secondary Efficacy Outcome - Composite of Death, MI, Stroke, HF, A. Revasc, or Angina. | 3-5 years
  The composite of cardiovascular death, myocardial infarction, stroke, heart failure, arterial revascularization, or unstable, new or worsening angina.
Secondary Efficacy Outcome - Event Outcome - CV Death | 3-5 years
  Cardiovascular death.
Secondary Efficacy Outcome - Event Outcome - Myocardial Infarction | 3-5 years
  Myocardial infarction.
Secondary Efficacy Outcome - Event Outcome - Stroke | 3-5 years
  Stroke.
Secondary Efficacy Outcome - Event Outcome - Heart Failure | 3-5 years
  Heart failure.
Secondary Efficacy Outcome - Event Outcome - Venous Thromboembolism | 3-5 years
  Venous Thromboembolism.

OTHER OUTCOMES:
Tertiary Efficacy Outcomes - Event Outcome - New or Worsening Angina | 3-5 years.
  New or worsening angina.
Tertiary Efficacy Outcomes - Event Outcome - New Atrial Fibrillation | 3-5 years
  New atrial fibrillation.
Tertiary Efficacy Outcomes - Cognitive Function | 3-5 years
  Cognitive function, as measured by the DSS test.
Tertiary Efficacy Outcomes - Physical Measurement - Grip Strength | 3-5 years
  Handgrip strength, as measured using the JAMAR Dynamometer.
Tertiary Efficacy Outcomes - Physical Measurement - Timed Walk Test | 3-5 years
  Timed-get-up-and-go-test.
Tertiary Efficacy Outcomes - Physical Measurement - Walk Test | 3-5 years
  Six-minute walk distance.
Tertiary Efficacy Outcomes - Physical Frailty | 3-5 years
  Physical Frailty
Tertiary Efficacy Outcomes - Physical Measurement - Waist | 3-5 years
  Waist circumference.
Tertiary Efficacy Outcomes - HbA1c | 3-5 years
  HbA1c concentration.
Tertiary Efficacy Outcomes - Lipid Profile | 3-5 years
  Lipid profile.
Tertiary Efficacy Outcomes - Event Outcome - Prostate Cancer Death | 3-5 years
  Prostate cancer death.
Tertiary Efficacy Outcomes - Prostate Cancer Characteristics - PC Progression | 3-5 years
  Distant prostate cancer progression.
Tertiary Efficacy Outcomes - Prostate Cancer Characteristics - Castrate-Resistant PC | 3-5 years
  Development of castrate-resistant prostate cancer
Tertiary Efficacy Outcomes - Prostate Cancer Characteristics - PSA Progression | 3-5 years
  PSA progression.
Tertiary Efficacy Outcomes - Prostate Cancer Characteristics - Biochemical Failure | 3-5 years
  Biochemical failure.
Safety Outcome - Emergent Adverse Event - Major Bleeding | 3-5 years
  Major bleeding.
Safety Outcome - Emergent Adverse Event - Myositis | 3-5 years
  Myositis.
Safety Outcome - Emergent Adverse Event - Liver Injury | 3-5 years
  Liver injury.
Safety Outcome - Emergent Adverse Event - Kidney Injury | 3-5 years
  Kidney injury.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Darryl Leong, MBBs,MPH,PhD,FRACP,FESC, Study Director — McMaster University
Locations (54):
- United States (2):
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - University of Kansas Medical Center, Kansas City, Kansas
- Australia (3):
  - Westmead Hospital, Westmead, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Center, Adelaide, South Australia
- Brazil (25):
  - Centro de Pesquisa Clínica do Brasil, Brasília, Federal District
  - Hospital Felício Rocho, Belo Horizonte, Minas Gerais
  - Universidade Federal do Triângulo Mineiro, Uberaba, Minas Gerais
  - Sociedade Hospitalar Angelina Caron, Campina Grande do Sul, Paraná
  - Nucleo de Pesquisa Clinica Hospital do Rocio, Campo Largo, Paraná
  - Centro Médico São Francisco, Curitiba, Paraná
  - Instituto De Medicina Integral Prof. Fernando Figueira - IMIP, Recife, Pernambuco
  - Instituto Nacional de Cardiologia, Rio de Janeiro, Rio de Janeiro
  - Hospital de Caridade de Ijuí, Ijuí, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Irmandade Da Santa Casa De Misericórdia De Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Mae de Deus, Porto Alegre, Rio Grande do Sul
  - Hospital Municipal de Barueri, Barueri, São Paulo
  - Faculdade de Medicina da Universidade Estadual Paulista - Campus de Botucatu - UNESP, Botucatu, São Paulo
  - Hospital Universitário São Francisco na Providência de Deus, Bragança Paulista, São Paulo
  - Fundacao Doutor Amaral Carvalho, Jaú, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto, São Paulo
  - Santa Casa de São Paulo (IPITEC), São Paulo, São Paulo
  - Hospital Alemao Oswaldo Cruz, São Paulo, São Paulo
  - Beneficência Nipo-Brasileira de São Paulo. Hospital Nipo-Brasileiro, São Paulo, São Paulo
  - Marina Leonardo, São Paulo, São Paulo
  - Instituto do Coração do Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo and Fundação Zerbini (Incor), São Paulo, São Paulo
  - Hospital Santa Marcelina, São Paulo, São Paulo
  - Instituto D'Or de Pesquisa e Ensino, São Paulo, São Paulo
  - Integral Pesquisa e Ensino, Votuporanga, São Paulo
- Canada (17):
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Queen's University, Kingston, Ontario
  - Grand River Hospital, Grand River Regional Cancer Centre, Kitchener, Ontario
  - London Health Sciences Centre, London, Ontario
  - London Health Sciences, Victoria Hospital, London, Ontario
  - Niagara Health, St. Catharines Site, Niagara, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network, Princess Margaret Cancer Centre, Toronto, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - University Hospital of Montreal, Montreal, Quebec
  - McGill University, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Laval University, Québec, Quebec
  - Centre Universitaire de Sherbrooke, Sherbrooke, Quebec
- Colombia (3):
  - Hospital Universitario San Ignacio, Bogotá, Cundinamarca
  - FOSCAL, Floridablanca, Santander Department
  - Fundacio Valle de Lili, Cali, Valle del Cauca Department
- Israel (3):
  - Heart Institute - Holon Medical Center, Holon
  - Rabin Medical Center, Petah Tikva
  - Tel-Aviv Sourasky Medical Centre, Tel Aviv
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dahan J, Pinthus J, Delouya G, Taussky D, Duceppe E, de Jesus A, Leong D. Investigation of association between clinically significant prostate cancer, obesity and platelet to-lymphocyte ratio and neutrophil -to-lymphocyte ratio. BMC Urol. 2024 Oct 16;24(1):226. doi: 10.1186/s12894-024-01617-2. PMID 39407194
- [Derived] Savija N, Leong DP, Pinthus J, Karampatos S, Shayegan B, Mian R, Rangarajan S, Fradet V, de Souza RJ, Mente A, Dehghan M. Development and Comparability of a Short Food-Frequency Questionnaire to Assess Diet in Prostate Cancer Patients: The Role of Androgen Deprivation Therapy in CArdiovascular Disease - A Longitudinal Prostate Cancer Study (RADICAL PC) Substudy. Curr Dev Nutr. 2021 Aug 12;5(11):nzab106. doi: 10.1093/cdn/nzab106. eCollection 2021 Nov. PMID 34870071